CLINICAL TRIAL: NCT01784679
Title: GNE-Myopathy Disease Monitoring Program (GNEM-DMP): A Registry and Prospective Observational Natural History Study to Assess GNE Myopathy or Hereditary Inclusion Body Myopathy (HIBM)
Status: Completed | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Other Study IDs: UX001-CL401
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Hereditary Inclusion Body Myopathy; GNE Myopathy; Nonaka Disease; Quadriceps Sparing Myopathy (QSM); Distal Myopathy With Rimmed Vacuoles (DMRV)
Keywords: Hereditary Inclusion Body Myopathy; GNE Myopathy; Nonaka Disease; Quadriceps Sparing Myopathy; distal myopathy with rimmed vacuoles; ultragenyx; rare disease
MeSH Terms: conditions — Distal myopathy, Nonaka type; Rare Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Natural History Prospective Observational Group
- Online Registry Patient Reported Group

SUMMARY:
HIBM is a severe progressive myopathy that typically presents in early adulthood as weakness in the distal muscles of the lower extremities and progresses proximally, leading to a loss of muscle strength and function, and ultimately a wheelchair-bound state. The rate of progression is gradual and variable over the course of 10-20 years or longer. There is a need to better understand the disease-specific features of HIBM to heighten disease awareness; facilitate early diagnosis; identify patients; expand knowledge of the clinical presentation, progression and variation of the disease; identify and validate biomarkers and other efficacy measures; inform on the design and interpretation of clinical studies of investigational products; and eventually to optimize patient management.

DETAILED DESCRIPTION:
The main objective of this program is to better understand HIBM.

The specific HIBM Disease Registry's objectives are to:

* Understand the geographic distribution and regional incidence/prevalence of GNEM.
* Obtain an assessment of the medical history, clinical presentation and progression of disease in GNEM patients and provide a connection for subjects to the broader GNEM community and associated programs.
* Provide customized information to subjects and their physicians that desire information on their disease status and progression.

The specific HIBM Natural History Study's objectives are to:

* Characterize HIBM disease presentation and progression over time using relevant clinical assessments of muscle strength and function.
* Obtain information to better characterize quality of life and understand the timing of significant life changing events in HIBM patients using patient-reported outcomes.
* Identify biomarkers and efficacy measures for use as endpoints in future clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing and able to provide electronic consent to release access to medical information to the study sponsor or its agents
* Must have a diagnosis of GNEM, HIBM, Quadriceps Sparing Myopathy (QSM), Inclusion Body Myopathy Type 2, distal myopathy with rimmed vacuoles (DMRV), or Nonaka disease. (Genotyping will not be required for the GNEM Disease Registry and will not be conducted in this protocol. However, when available, genotypes of disease registry subjects should be provided and all subjects will be encouraged to be genotyped during the course of the disease registry through independent programs.)
* Must be willing and able to comply with all study procedures.
* Must meet all of the inclusion criteria for the GNEM Disease Registry portion of the study.
* Must be willing to have their collected information used as part of the GNEM Disease Registry.
* Must provide a genotype confirming GNE disease. Genotyping will not be conducted as part of this protocol, so GNE disease genotype data must be provided by the subject/physician from other sources.
* In the opinion of the investigator, the subject will be complaint with study visit schedule and study procedures.

Exclusion Criteria:

* For Natural History Component, concurrent disease or condition that, in the view of the investigator, would interfere with study participation or would affect safety.
* For Online Registry Component, there are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Must have a diagnosis of HIBM, GNE myopathy, Quadriceps Sparing Myopathy (QSM), Inclusion Body Myopathy Type 2, distal myopathy with rimmed vacuoles (DMRV), or Nonaka disease.
Sampling Method: Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2013-04-05 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Characterize HIBM disease presentation and progression over time using relevant clinical assessments of muscle strength and function. | 3 years

SECONDARY OUTCOMES:
Obtain information to better characterize quality of life and understand the timing of significant life changing events in HIBM patients using patient-reported outcomes. | 3 years

CONTACTS AND LOCATIONS:
Locations (5):
- University of California, Irvine, Irvine, California, United States
- Bulgarian Neuromuscular Disease Association, Sofia, Bulgaria
- McMaster University, Hamilton, Ontario, Canada
- Association Institut de Myologie, Paris, France
- The Newcastle upon Tyne Hospitals, Newcastle upon Tyne, Tyne and Wear, United Kingdom